CLINICAL TRIAL: NCT00305162
Title: A Clinical Trial Comparing Cangrelor to Clopidogrel in Subjects Who Require Percutaneous Coronary Intervention (PCI).
Brief Title: A Clinical Trial to Demonstrate the Efficacy of Cangrelor
Acronym: PCI
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient evidence of the clinical effectiveness of cangrelor
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TMC-CAN-05-02
Record Dates: First submitted 2006-03-17; First posted 2006-03-21 (Estimated); Results first posted 2014-04-23 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Myocardial Infarction (MI); Acute Coronary Syndromes (ACS)
Keywords: Acute Coronary Syndrome (ACS); Percutaneous Coronary Intervention (PCI); non-ST-segment elevation myocardial infarction (NSTEMI); ST-segment elevation myocardial infarction (STEMI)
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome; Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction | interventions — cangrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cangrelor (Experimental): placebo capsules (to match) + cangrelor bolus (30 mcg/kg) & infusion (4 mcg/kg/min) administered from randomization for at least 2 hours, or until the end of the PCI, whichever is longer with the option to extend up to 4 hours maximum (per investigator discretion) + active clopidogrel (600mg) post infusion
  Interventions: Drug: Cangrelor (P2Y12 inhibitor); Drug: clopidogrel (oral P2Y12 inhibitor); Drug: Placebo capsules - as soon as possible after randomization
- Clopidogrel (Active Comparator): clopidogrel capsules (600 mg) + placebo bolus & infusion (to match) + placebo capsules (to match) post infusion
  Interventions: Drug: clopidogrel (oral P2Y12 inhibitor); Drug: Placebo bolus & placebo infusion; Drug: Placebo capsules - end of infusion

INTERVENTIONS:
Drug: Cangrelor (P2Y12 inhibitor) — IV bolus (30 mcg/kg) & infusion (4 mcg/kg/min) initiated prior to PCI, as soon as possible following randomization (after need for PCI is confirmed) but not more than 30 minutes prior to placement of arterial access. Infusion is to continue for at least 2 hours, or until the end of the PCI, whichever is longer with the option to extend up to 4 hours maximum (per investigator discretion).
  Arms: Cangrelor
Drug: clopidogrel (oral P2Y12 inhibitor) — 600 mg active clopidogrel administered as soon as possible following randomization (after need for PCI confirmed), but not more than 30 minutes prior to the placement of the arterial access.
  Other Names: Plavix
Drug: Placebo bolus & placebo infusion — placebo bolus (30 mcg/kg) & placebo infusion (4 mcg/kg/min) administered from randomization for at least 2 hours, or until the end of the PCI, whichever is longer with the option to extend up to 4 hours maximum (per investigator discretion)
  Arms: Clopidogrel
Drug: Placebo capsules - end of infusion — Placebo capsules given at the end of infusion to mimic 600mg clopidogrel dosing
  Arms: Clopidogrel
Drug: Placebo capsules - as soon as possible after randomization — Placebo capsules given as soon as possible after randomization to mimic 600mg clopidogrel dosing
  Arms: Cangrelor

SUMMARY:
The primary objective of this study is to demonstrate that the efficacy of cangrelor is superior, or at least non-inferior, to that of clopidogrel in subjects requiring PCI.

ELIGIBILITY:
INCLUSION CRITERIA

To be included in this study, subjects must meet the following criteria:

* Angiography demonstrating atherosclerosis amenable to treatment by percutaneous coronary intervention (PCI) with or without stent implantation and diagnosis of Acute Coronary Syndrome (ACS) by elevated cardiac markers or ischemic chest discomfort w/electrocardiogram changes + age > 65 or diabetes or ST-elevation MI.

EXCLUSION CRITERIA

Subjects will be excluded from the study if they present with any of the following:

1. Not a candidate for PCI
2. Increased bleeding risk: ischemic stroke within the last year or any previous hemorrhagic stroke, tumor, cerebral arteriovenous malformation, or intracranial aneurysm; recent (<1 month) trauma or major surgery (including by-pass surgery); currently receiving warfarin, active bleeding
3. Impaired hemostasis: known International Normalized Ratio (INR) >1.5 at screening; past or present bleeding disorder (including congenital bleeding disorders such as von Willebrand's disease or hemophilia, acquired bleeding disorders, and unexplained clinically significant bleeding disorders), thrombocytopenia (platelet count <100,000/µL), or history of thrombocytopenia or neutropenia associated with clopidogrel
4. Severe hypertension not adequately controlled by antihypertensive therapy at the time of randomization
5. Receipt of fibrinolytic therapy in the 12 hours preceding randomization
6. Receipt of clopidogrel dose exceeding maintenance dose (ie, >75 mg) at any time in the 5 days preceding randomization
7. Inability to swallow study capsules
8. Glycoprotein IIb/IIIa (GPI) Inhibitor usage within the previous 12 hours [applicable to unstable angina (UA) and non-ST-elevation myocardial infarction (NSTEMI) patients]

Subjects excluded for any of the above reasons may be re-screened for participation at any time if the exclusion characteristic has changed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8882 (Actual)
Dates: Start 2006-04; Primary Completion 2009-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepak L. Bhatt, MD, Principal Investigator — The Cleveland Clinic; Robert A. Harrington, MD, Principal Investigator — Duke University Medical Center and Duke Clinical Research Institute; Simona Skerjanec, PharmD, Study Director — The Medicines Company
Locations (1):
- Pennsylvania Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Harrington RA, Stone GW, McNulty S, White HD, Lincoff AM, Gibson CM, Pollack CV Jr, Montalescot G, Mahaffey KW, Kleiman NS, Goodman SG, Amine M, Angiolillo DJ, Becker RC, Chew DP, French WJ, Leisch F, Parikh KH, Skerjanec S, Bhatt DL. Platelet inhibition with cangrelor in patients undergoing PCI. N Engl J Med. 2009 Dec 10;361(24):2318-29. doi: 10.1056/NEJMoa0908628. PMID 19915221
- [Derived] Gutierrez JA, Harrington RA, Stone GW, Steg PG, Gibson CM, Hamm CW, Price MJ, Lopes RD, Leonardi S, Prats J, Deliargyris EN, Mahaffey KW, White HD, Bhatt DL; CHAMPION Investigators. Efficacy and safety of cangrelor in patients with peripheral artery disease undergoing percutaneous coronary intervention - Insights from the CHAMPION program. Am Heart J Plus. 2021 Aug 25;9:100043. doi: 10.1016/j.ahjo.2021.100043. eCollection 2021 Sep. PMID 38551015
- [Derived] Peterson BE, Harrington RA, Stone GW, Steg PG, Gibson CM, Hamm CW, Price MJ, Lopes RD, Leonardi S, Prats J, Deliargyris EN, Mahaffey KW, White HD, Bhatt DL. Effect of Platelet Inhibition by Cangrelor Among Obese Patients Undergoing Coronary Stenting: Insights From CHAMPION. Circ Cardiovasc Interv. 2022 Mar;15(3):e011069. doi: 10.1161/CIRCINTERVENTIONS.121.011069. Epub 2022 Feb 24. PMID 35196863
- [Derived] Groves EM, Bhatt DL, Steg PG, Deliargyris EN, Stone GW, Gibson CM, Hamm CW, Mahaffey KW, White HD, Angiolillo DJ, Prats J, Harrington RA, Price MJ. Incidence, Predictors, and Outcomes of Acquired Thrombocytopenia After Percutaneous Coronary Intervention: A Pooled, Patient-Level Analysis of the CHAMPION Trials (Cangrelor Versus Standard Therapy to Achieve Optimal Management of Platelet Inhibition). Circ Cardiovasc Interv. 2018 Apr;11(4):e005635. doi: 10.1161/CIRCINTERVENTIONS.117.005635. PMID 29632238
- [Derived] Vaduganathan M, Harrington RA, Stone GW, Steg G, Gibson CM, Hamm CW, Price MJ, Lopes RD, Leonardi S, Deliargyris EN, Prats J, Mahaffey KW, White HD, Bhatt DL. Short- and long-term mortality following bleeding events in patients undergoing percutaneous coronary intervention: insights from four validated bleeding scales in the CHAMPION trials. EuroIntervention. 2018 Feb 2;13(15):e1841-e1849. doi: 10.4244/EIJ-D-17-00723. PMID 28988157
- [Derived] Parker WA, Bhatt DL, Prats J, Day JRS, Steg PG, Stone GW, Hamm CW, Mahaffey KW, Price MJ, Gibson CM, White HD, Storey RF; CHAMPION PHOENIX Investigators. Characteristics of dyspnoea and associated clinical outcomes in the CHAMPION PHOENIX study. Thromb Haemost. 2017 Jun 2;117(6):1093-1100. doi: 10.1160/TH16-12-0958. Epub 2017 Apr 6. PMID 28382371
- [Derived] Vaduganathan M, Harrington RA, Stone GW, Deliargyris EN, Steg PG, Gibson CM, Hamm CW, Price MJ, Menozzi A, Prats J, Elkin S, Mahaffey KW, White HD, Bhatt DL. Evaluation of Ischemic and Bleeding Risks Associated With 2 Parenteral Antiplatelet Strategies Comparing Cangrelor With Glycoprotein IIb/IIIa Inhibitors: An Exploratory Analysis From the CHAMPION Trials. JAMA Cardiol. 2017 Feb 1;2(2):127-135. doi: 10.1001/jamacardio.2016.4556. PMID 27902833
- [Derived] White HD, Chew DP, Dauerman HL, Mahaffey KW, Gibson CM, Stone GW, Gruberg L, Harrington RA, Bhatt DL. Reduced immediate ischemic events with cangrelor in PCI: a pooled analysis of the CHAMPION trials using the universal definition of myocardial infarction. Am Heart J. 2012 Feb;163(2):182-90.e4. doi: 10.1016/j.ahj.2011.11.001. PMID 22305835

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were selected for randomization based on the need for percutaneous coronary intervention (PCI). Randomization could only occur after the need for PCI was confirmed by angiography, with the exception of ST-segment elevation myocardial infarction (STEMI) patients, who could be enrolled upon confirmation of STEMI by electrocardiogram (ECG).
Groups:
- Cangrelor Arm: cangrelor arm: placebo capsules at PCI start + cangrelor bolus(30 mcg/kg) & infusion (4mcg/kg/min) followed by clopidogrel (600 mg) post infusion
- Clopidogrel Arm: clopidogrel arm: clopidogrel capsules (600 mg)at PCI start + placebo bolus & infusion followed by placebo capsules post infusion
Period: 48 Hour Follow-up Period
Arm/Group | Cangrelor Arm | Clopidogrel Arm
Started | 4435 | 4447
Intent-to-treat (ITT): SA/UA/NSTEMI | 3933 (Patients who completed through 48 hours) | 3924 (Patients who completed through 48 hours)
Intent-to-treat (ITT): STEMI | 482 (Patients who completed through 48 hours) | 507 (Patients who completed through 48 hours)
Modified ITT (mITT): SA/UA/NSTEMI | 3889 (Completed through 48 hours; Excludes those who did not receive study drug or undergo index PCI.) | 3865 (Completed through 48 hours; Excludes those who did not receive study drug or undergo index PCI.)
Modified ITT (mITT): STEMI | 446 (Completed through 48 hours; Excludes those who did not receive study drug or undergo index PCI.) | 447 (Completed through 48 hours; Excludes those who did not receive study drug or undergo index PCI.)
Safety Population | 4374 (Patients who received at least 1 dose of study drug, according to the actual treatment received.) | 4365 (Patients who received at least 1 dose of study drug, according to the actual treatment received.)
Completed | 4415 (intent-to-treat (ITT) completers at 48 hour follow-up) | 4431 (intent-to-treat (ITT) completers at 48 hour follow-up)
Not Completed | 20 | 16
Period: 30-day Follow-up Period
Arm/Group | Cangrelor Arm | Clopidogrel Arm
Started | 4435 | 4447
Intent-to-treat (ITT): SA/UA/NSTEMI | 3902 (Completed through 30-days) | 3883 (Completed through 30-days)
Intent-to-treat (ITT): STEMI | 471 (Completed through 30-days) | 501 (Completed through 30-days)
Modified ITT (mITT): SA/UA/NSTEMI | 3860 (Completed through 30-days; Excludes those who did not receive study drug or undergo index PCI.) | 3827 (Completed through 30-days; Excludes those who did not receive study drug or undergo index PCI.)
Modified ITT (mITT): STEMI | 438 (Completed through 30-days; Excludes those who did not receive study drug or undergo index PCI.) | 444 (Completed through 30-days; Excludes those who did not receive study drug or undergo index PCI.)
Completed | 4373 (intent-to-treat (ITT) completers at 30-day follow-up) | 4384 (intent-to-treat (ITT) completers at 30-day follow-up)
Not Completed | 62 | 63
Period: 1 Year Follow-up Period
Arm/Group | Cangrelor Arm | Clopidogrel Arm
Started | 4435 | 4447
Intent-to-treat (ITT): SA/UA/NSTEMI | 3900 (Completed through 1 year) | 3878 (Completed through 1 year)
Intent-to-treat (ITT): STEMI | 480 (Completed through 1 year) | 504 (Completed through 1 year)
Modified ITT (mITT): SA/UA/NSTEMI | 3851 (Completed through 1 year; Excludes those who did not receive study drug or undergo index PCI.) | 3818 (Completed through 1 year; Excludes those who did not receive study drug or undergo index PCI.)
Modified ITT (mITT): STEMI | 446 (Completed through 1 year; Excludes those who did not receive study drug or undergo index PCI.) | 444 (Completed through 1 year; Excludes those who did not receive study drug or undergo index PCI.)
Completed | 4380 (intent-to-treat (ITT) completers at 1-year follow-up) | 4382 (intent-to-treat (ITT) completers at 1-year follow-up)
Not Completed | 55 | 65

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population
Groups:
- Cangrelor Arm: cangrelor arm: placebo capsules (to match) at PCI start + cangrelor bolus (30 mcg/kg) & infusion (4mcg/kg/min) followed by clopidogrel (600 mg) post infusion
- Clopidogrel Arm: clopidogrel arm: clopidogrel capsules (600 mg) at PCI start + placebo bolus & infusion (to match) followed by placebo capsules post infusion
- Total: Total of all reporting groups
Arm/Group | Cangrelor Arm | Clopidogrel Arm | Total
Number analyzed (Participants) | 4433 | 4444 | 8877
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (11.3) | 62.2 (11.5) | 62.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1158 | 1235 | 2393
  Male | 3275 | 3209 | 6484
Region of Enrollment [Number; unit: participants]
  United States | 2629 | 2638 | 5267
  Australia | 233 | 237 | 470
  Argentina | 25 | 26 | 51
  Austria | 215 | 215 | 430
  Brazil | 111 | 116 | 227
  Canada | 10 | 5 | 15
  Georgia | 228 | 230 | 458
  Germany | 162 | 156 | 318
  India | 260 | 260 | 520
  Italy | 169 | 167 | 336
  New Zealand | 110 | 116 | 226
  Poland | 231 | 232 | 463
  Spain | 11 | 7 | 18
  Ukraine | 39 | 39 | 78

OUTCOME MEASURES:

1. Primary Outcome: Incidence of All-cause Mortality, Myocardial Infarction (MI), and Ischemia-driven Revascularization (IDR)
Description: (composite incidence)
Time Frame: randomization through 48 hours after randomization
Population: mITT (excluding STEMI)
Measure: Number; unit: participants
Groups:
- Cangrelor Arm: placebo capsules (to match) at PCI start + cangrelor bolus (30 mcg/kg) & infusion (4 mcg/kg/min) administered from randomization for at least 2 hours, or until the end of the PCI, whichever is longer with the option to extend up to 4 hours maximum (per investigator discretion) + active clopidogrel (600mg) post infusion
- Clopidogrel Arm: clopidogrel capsules (600 mg)at PCI start + placebo bolus & infusion (to match) followed by placebo capsules post infusion
Arm/Group | Cangrelor Arm | Clopidogrel Arm
Number analyzed (Participants) | 3889 | 3865
participants | 290 [0.89 to 1.24] | 276 [0.98 to 1.24]

2. Secondary Outcome: Incidence of All-cause Mortality and MI
Description: (composite incidence)
Time Frame: randomization through 48 hours after randomization
Population: mITT (excluding STEMI)
Measure: Number; unit: participants
Groups:
- Clopidogrel Arm: clopidogrel capsules (600 mg) at PCI start + placebo bolus & infusion (to match) followed by placebo capsules post infusion
Arm/Group | Cangrelor Arm | Clopidogrel Arm
Number analyzed (Participants) | 3889 | 3865
participants | 285 | 261

3. Secondary Outcome: Individual Incidence of All-cause Mortality
Time Frame: randomization through 48 hours after randomization
Population: mITT (excluding STEMI)
Measure: Number; unit: participants
Arm/Group | Cangrelor Arm | Clopidogrel Arm
Number analyzed (Participants) | 3889 | 3865
participants | 8 | 5

4. Secondary Outcome: Individual Incidence of IDR
Time Frame: randomization through 48 hours after randomization
Population: mITT (excluding STEMI)
Measure: Number; unit: participants
Arm/Group | Cangrelor Arm | Clopidogrel Arm
Number analyzed (Participants) | 3889 | 3865
participants | 13 | 23

5. Secondary Outcome: Incidence of Stroke
Description: Stroke is defined as a sudden, focal neurological defect resulting from a cerebrovascular cause that is not reversible within 24 hours and not due to a readily identifiable cause such as a tumor or trauma. All suspected strokes were reviewed and adjudicated by the Clinical Events Committee (CEC) who considered all clinically relevant information and imaging studies to classify all strokes as:
  * primary hemorrhagic - stroke with focal collections of intracranial blood
  * ischemic cerebral infarction - stroke without focal collections of intracranial blood
  * infarction with hemorrhagic conversion - cerebral infarction with blood thought to represent hemorrhagic conversion and not primary bleeding
  * uncertain - no imaging or autopsy data are available.
Time Frame: randomization through 48 hours after randomization
Population: mITT (excluding STEMI)
Measure: Number; unit: participants
Arm/Group | Cangrelor Arm | Clopidogrel Arm
Number analyzed (Participants) | 3889 | 3865
participants
  primary hemorrhagic | 1 | 0
  infarction with hemorrhagic conversion | 0 | 0
  cerebral infarction | 5 | 7
  uncertain type | 0 | 0

6. Secondary Outcome: Incidence of Abrupt Closure, Threatened Abrupt Closure, Need for Urgent Coronary Artery Bypass Graft (CABG) Surgery, or Unsuccessful Procedure During the Index PCI
Description: (a patient could have multiple procedural events)
Time Frame: during index PCI
Population: mITT (excluding STEMI) and based on available data
Measure: Number; unit: participants
Arm/Group | Cangrelor Arm | Clopidogrel Arm
Number analyzed (Participants) | 3897 | 3871
participants | 127 | 141

7. Secondary Outcome: Incidence of All-cause Mortality, MI or IDR
Description: (composite incidence)
Time Frame: randomization through 30 days after randomization
Population: mITT (excluding STEMI), based on 30-day completers
Measure: Number; unit: participants
Arm/Group | Cangrelor Arm | Clopidogrel Arm
Number analyzed (Participants) | 3860 | 3827
participants | 343 | 327

8. Secondary Outcome: Incidence of All-cause Mortality or MI
Description: (composite incidence)
Time Frame: randomization through 30 days after randomization
Population: mITT (excluding STEMI), based on 30-day completers
Measure: Number; unit: participants
Arm/Group | Cangrelor Arm | Clopidogrel Arm
Number analyzed (Participants) | 3860 | 3827
participants | 321 | 298

9. Secondary Outcome: Incidence of All-cause Mortality
Time Frame: randomization through 30 days after randomization
Population: mITT (excluding STEMI), based on 30-day completers
Measure: Number; unit: participants
Arm/Group | Cangrelor Arm | Clopidogrel Arm
Number analyzed (Participants) | 3860 | 3827
participants | 34 | 29

10. Secondary Outcome: Incidence of MI
Time Frame: randomization through 30 days after randomization
Population: mITT (excluding STEMI), based on 30-day completers
Measure: Number; unit: participants
Arm/Group | Cangrelor Arm | Clopidogrel Arm
Number analyzed (Participants) | 3860 | 3827
participants | 297 | 276

11. Secondary Outcome: Incidence of IDR
Time Frame: randomization through 30 days after randomization
Population: mITT (excluding STEMI), based on 30-day completers
Measure: Number; unit: participants
Arm/Group | Cangrelor Arm | Clopidogrel Arm
Number analyzed (Participants) | 3860 | 3827
participants | 44 | 52

12. Secondary Outcome: Incidence of Stroke
Time Frame: randomization through 30 days after randomization
Population: mITT (excluding STEMI), based on available data
Measure: Number; unit: participants
Arm/Group | Cangrelor Arm | Clopidogrel Arm
Number analyzed (Participants) | 3860 | 3827
participants | 5 | 7

13. Secondary Outcome: Incidence of All Cause Mortality
Description: (excluding STEMI)
Time Frame: randomization through 1 year after randomization
Population: mITT (excluding STEMI), based on 1 year completers
Measure: Number; unit: participants
Arm/Group | Cangrelor Arm | Clopidogrel Arm
Number analyzed (Participants) | 3851 | 3818
participants | 116 [0.75 to 1.20] | 120 [0.75 to 1.20]

14. Secondary Outcome: Incidence of GUSTO Severe / Life-threatening Bleeding
Description: Major bleeding (non-CABG-related) - Safety population
Time Frame: randomization through 48 hours after randomization
Population: Safety Population (inclusive of STEMI patients)
Measure: Number; unit: participants
Arm/Group | Cangrelor Arm | Clopidogrel Arm
Number analyzed (Participants) | 4374 | 4365
participants | 10 | 11

15. Secondary Outcome: Incidence of Thrombolysis in Myocardial Infarction (TIMI) Major Bleeding
Description: Major bleeding (non-CABG-related) - Safety population
Time Frame: randomization through 48 hours after randomization
Population: Safety Population (inclusive of STEMI patients)
Measure: Number; unit: participants
Arm/Group | Cangrelor Arm | Clopidogrel Arm
Number analyzed (Participants) | 4374 | 4365
participants | 19 | 14

16. Secondary Outcome: Incidence of ACUITY Major Bleeding
Description: Major bleeding (non-CABG-related) - Safety population
Time Frame: randomization through 48 hours after randomization
Population: Safety Population (inclusive of STEMI patients)
Measure: Number; unit: participants
Arm/Group | Cangrelor Arm | Clopidogrel Arm
Number analyzed (Participants) | 4374 | 4365
participants | 151 | 120

17. Secondary Outcome: Incidence of ACUITY Major Bleeding (Without Hematoma >/= 5 cm)
Description: excludes ACUITY major bleeding for which the only qualifying event was hematoma >/= 5 cm
Time Frame: randomization through 48 hours after randomization
Population: Safety Population (inclusive of STEMI patients)
Measure: Number; unit: participants
Arm/Group | Cangrelor Arm | Clopidogrel Arm
Number analyzed (Participants) | 4374 | 4365
participants | 78 | 65

ADVERSE EVENTS:
Groups:
- Clopidogrel Arm: clopidogrel arm: clopidogrel capsules (600 mg)at PCI start + placebo bolus & infusion (to match) followed by placebo capsules post infusion
Arm/Group | Cangrelor Arm | Clopidogrel Arm
Serious Adverse Events (participants affected / at risk) | 125/4374 | 127/4365
Other Adverse Events (participants affected / at risk) | 1149/4374 | 1159/4365
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cangrelor Arm (N=4374) | Clopidogrel Arm (N=4365)
anaemia (Blood and lymphatic system disorders) | 1 | 0
haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 2
leukocytosis (Blood and lymphatic system disorders) | 0 | 1
thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
acute myocardial infarction (Cardiac disorders) | 1 | 0
angina pectoris (Cardiac disorders) | 4 | 3
arrhythmia (Cardiac disorders) | 0 | 1
arrhythmia supraventricular (Cardiac disorders) | 0 | 1
arteriospasm coronary (Cardiac disorders) | 1 | 0
atrial fibrillation (Cardiac disorders) | 2 | 2
atrial flutter (Cardiac disorders) | 0 | 1
atrial tachycardia (Cardiac disorders) | 0 | 1
atrioventricular block (Cardiac disorders) | 0 | 1
atrioventricular block third degree (Cardiac disorders) | 2 | 2
bradycardia (Cardiac disorders) | 2 | 3
cardiac arrest (Cardiac disorders) | 4 | 6
cardiac failure (Cardiac disorders) | 2 | 0
cardiac failure acute (Cardiac disorders) | 1 | 1
cardiac failure congestive (Cardiac disorders) | 4 | 3
cardiac tamponade (Cardiac disorders) | 1 | 0
cardiogenic shock (Cardiac disorders) | 6 | 8
coronary artery dissection (Cardiac disorders) | 5 | 3
coronary artery occlusion (Cardiac disorders) | 0 | 3
coronary artery perforation (Cardiac disorders) | 4 | 2
coronary artery thrombosis (Cardiac disorders) | 1 | 0
in-stent arterial restenosis (Cardiac disorders) | 0 | 1
myocardial infarction (Cardiac disorders) | 0 | 1
nodal rhythm (Cardiac disorders) | 1 | 0
pericardial effusion (Cardiac disorders) | 1 | 0
sick sinus syndrome (Cardiac disorders) | 3 | 0
sinus arrest (Cardiac disorders) | 0 | 2
supraventricular tachycardia (Cardiac disorders) | 0 | 1
ventricular arrhythmia (Cardiac disorders) | 1 | 0
ventricular asystole (Cardiac disorders) | 1 | 0
ventricular fibrillation (Cardiac disorders) | 12 | 6
ventricular tachycardia (Cardiac disorders) | 4 | 5
retinal artery occlusion (Eye disorders) | 1 | 0
abdominal pain upper (Gastrointestinal disorders) | 1 | 0
haematemesis (Gastrointestinal disorders) | 0 | 1
retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
vomiting (Gastrointestinal disorders) | 0 | 2
cardiac death (General disorders) | 1 | 0
chest discomfort (General disorders) | 0 | 1
chest pain (General disorders) | 7 | 9
non-cardiac chest pain (General disorders) | 2 | 1
puncture site haemorrhage (General disorders) | 0 | 1
pyrexia (General disorders) | 1 | 0
sudden cardiac death (General disorders) | 1 | 0
sudden death (General disorders) | 0 | 1
vessel puncture site haematoma (General disorders) | 1 | 0
cholecystitis acute (Hepatobiliary disorders) | 1 | 2
gallbladder disorder (Hepatobiliary disorders) | 0 | 1
bronchitis (Infections and infestations) | 0 | 1
bronchitis viral (Infections and infestations) | 0 | 1
cellulitis (Infections and infestations) | 2 | 0
haematoma infection (Infections and infestations) | 1 | 0
pneumonia (Infections and infestations) | 1 | 3
sepsis (Infections and infestations) | 0 | 1
urinary tract infection (Infections and infestations) | 3 | 0
fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
thrombosis in device (Injury, poisoning and procedural complications) | 1 | 3
vascular procedure complication (Injury, poisoning and procedural complications) | 0 | 1
aspartate aminotransferase increased (Investigations) | 0 | 1
cardiac enzymes increased (Investigations) | 0 | 1
liver function test abnormal (Investigations) | 1 | 0
gout (Metabolism and nutrition disorders) | 1 | 0
hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
cerebral haemorrhage (Nervous system disorders) | 1 | 0
diabetic neuropathy (Nervous system disorders) | 0 | 1
presyncope (Nervous system disorders) | 2 | 2
syncope (Nervous system disorders) | 1 | 1
alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
depression (Psychiatric disorders) | 1 | 0
mental status changes (Psychiatric disorders) | 0 | 1
renal artery stenosis (Renal and urinary disorders) | 0 | 1
renal failure (Renal and urinary disorders) | 2 | 1
renal failure acute (Renal and urinary disorders) | 11 | 5
renal failure chronic (Renal and urinary disorders) | 0 | 2
acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 0
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 2
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2
angioneurotic oedema (Skin and subcutaneous tissue disorders) | 1 | 0
stent removal (Surgical and medical procedures) | 0 | 1
arterial thrombosis limb (Vascular disorders) | 1 | 1
artery dissection (Vascular disorders) | 0 | 1
embolism (Vascular disorders) | 1 | 0
femoral artery dissection (Vascular disorders) | 0 | 1
femoral artery occlusion (Vascular disorders) | 0 | 1
haemodynamic instability (Vascular disorders) | 0 | 1
hypertension (Vascular disorders) | 0 | 1
hypertensive emergency (Vascular disorders) | 0 | 2
hypotension (Vascular disorders) | 7 | 8
orthostatic hypotension (Vascular disorders) | 1 | 0
peripheral ischaemia (Vascular disorders) | 1 | 1
reperfusion injury (Vascular disorders) | 0 | 1
shock haemorrhagic (Vascular disorders) | 0 | 1
thrombosis (Vascular disorders) | 1 | 1
vascular pseudoaneurysm (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cangrelor Arm (N=4374) | Clopidogrel Arm (N=4365)
chest pain (General disorders) | 178 | 163
back pain (Musculoskeletal and connective tissue disorders) | 167 | 164
nausea (Gastrointestinal disorders) | 112 | 145
hypotension (Vascular disorders) | 97 | 89
headache (Nervous system disorders) | 93 | 97
vomiting (Gastrointestinal disorders) | 70 | 78
puncture site pain (General disorders) | 67 | 52
pyrexia (General disorders) | 45 | 37
dyspnea (Respiratory, thoracic and mediastinal disorders) | 42 | 16
ventricular tachycardia (Cardiac disorders) | 37 | 35
hypertension (Vascular disorders) | 32 | 34
chest discomfort (General disorders) | 32 | 24
bradycardia (Cardiac disorders) | 29 | 35
atrial fibrillation (Cardiac disorders) | 27 | 18
angina pectoris (Cardiac disorders) | 20 | 34
pain in extremity (Musculoskeletal and connective tissue disorders) | 20 | 24
syncope vasovagal (Nervous system disorders) | 17 | 26
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 17 | 23
dizziness (Nervous system disorders) | 17 | 21
anxiety (Psychiatric disorders) | 16 | 22
dyspepsia (Gastrointestinal disorders) | 14 | 22

LIMITATIONS AND CAVEATS:
Discontinued per prespecified stopping rules after the 70% interim analyses was conducted indicating the trial was not likely to meet the goal of demonstrating superiority to clopidogrel administered as usual care. No safety issues were identified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI communications regarding trial results are prohibited until after the communication and publication of the multi-center results by Sponsor, but no more than 12 months after conclusion of the trial at all sites.

PI must submit results communications to sponsor for review at least 40 days prior to submission for publication and Sponsor may embargo such communications for a period that is less than or equal to 135 days solely to seek appropriate patent protection.